CLINICAL TRIAL: NCT04871386
Title: #Stayhealthy - Monitoring Und Erhalt Der Psychischen Gesundheit Unter Bedingungen Sozialer Isolation während Der Corona-Krise
Brief Title: #Stayhealthy - Monitoring and Maintenance of Mental Health Under Conditions of Social Isolation During the Corona Crisis
Acronym: stayhealthy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 228/2020BO2
Record Dates: First submitted 2021-01-28; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-01

CONDITIONS: Mental Health Wellness 1
Keywords: anxiety; stress; depression; COVID-19; Corona virus
MeSH Terms: conditions — Anxiety Disorders; Depression; COVID-19 | interventions — Exercise; Psychology, Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acceptance and commitment therapy (ACT) (Experimental): 14 consecutive days of exercises (prompted via email every morning) derived from acceptance and commitment therapy (ACT); the instructions were text-based, contained a brief introduction to the general goal and the exercise of the day; the exercises were designed to be completable individually in 20 minutes. Additionally: completion of a daily review questionnaire ("online diary") including two open questions (Relevant events during the day? Helpful things for coping positively with the current situation?)
  Interventions: Behavioral: Acceptance and commitment therapy (ACT) exercises
- Positive psychology intervention (PP) (Experimental): 14 consecutive days of exercises (prompted via email every morning) derived from positive psychology (PP) interventions; the instructions were text-based, contained a brief introduction to the general goal and the exercise of the day; the exercises were designed to be completable individually in 20 minutes. Additionally: completion of a daily review questionnaire ("online diary") including two open questions (Relevant events during the day? Helpful things for coping positively with the current situation?)
  Interventions: Behavioral: Positive psychology (PP) exercises
- Control group (No Intervention): completion of a daily review questionnaire ("online diary") including two open questions (Relevant events during the day? Helpful things for coping positively with the current situation?); no additional intervention

INTERVENTIONS:
Behavioral: Acceptance and commitment therapy (ACT) exercises — The ACT group received 14 (partially succeeding) daily exercises, with each of the following categories being focused twice: Acceptance, contact with the present moment, cognitive defusion, self as context, personal values and committed action. The exercises consisted of metaphors and questions for self-reflection, explanations about emotions and thoughts with techniques to handle them differently, as well as a body scan.
  Arms: Acceptance and commitment therapy (ACT)
Behavioral: Positive psychology (PP) exercises — The PP group received 14 daily exercises that were derived from positive psychology interventions that have been proven effective in alleviating clinical symptoms and increasing subjective well-being. In detail, these were: Identifying positive emotions and ways to increase them; Enhancing pleasure from daily activities; Writing a gratitude letter; Identifying and appreciating three personal traits; Receiving a letter of support from one's future self; Taking different perspectives on one's current situation; Envisioning a perfect day; Identifying energy boosters and drainers; Identifying 3 character strengths and using one in a new way; Life review: Writing a legacy; Identifying the positive relationships in one's life; Doing an act of kindness; Three good things; and Coping with failure.
  Arms: Positive psychology intervention (PP)

SUMMARY:
The COVID-19 pandemic has led to a global health crisis with, so far, over 21 million registered cases and more than 700.000 deaths worldwide. In order to slow down the rate of new infections, millions of people have been directed to stay at home, thereby accepting severe restrictions of social contact and personal freedom to move. With fear of infection and economical loss as additional burdens, the current conditions have led to a significant increase in psychological distress and risk for the onset of mental disorders among the general population. Empirical evidence on effective measures to support mental health in COVID-19 "homestayers" is lacking.

In the present study, the investigators therefore used a randomized controlled trial (RCT) design to investigate the effects of two online intervention programs derived either from the field of positive psychology (PP) or acceptance and commitment therapy (ACT) with a third group of participants writing an online diary only (control group). Furthermore, over the entire study period, individual daily coping strategies were collected. A total of 138 adult German "homestayers" participated in the RCT with two weeks of daily interventions during the first "lock-down" period in Germany (April 19th to May 3rd 2020). Measures of stress, mental health (depression, anxiety) and subjective well-being (subjective vitality, overall well-being) were collected at baseline, at the end of the two-week intervention period and another 14 days after that (follow-up).

DETAILED DESCRIPTION:
A total of 138 individuals - recruited via university-wide emails and social media - completed the baseline questionnaire and agreed to participate in the study. Inclusion criteria were an age between 18 and 70 years, knowledge of the German language as well as conditions of increased social isolation at the beginning of the study. The latter criterion was operationalized by only including individuals who were currently staying mostly at home due to the Corona crisis (home office; quarantine measures; stay-at-home orders) with no (or only very few) direct contacts outside of their own household. The only relevant exclusion criterion was an acute diagnosis (within the last 3 months) of a mental disorder by a medical professional.

Procedure: A link in the invitation email of the study led to the online platform SoSciSurvey, where participants received information about the study, standards of data security, gave informed consent to participate and filled out pre-measures (t1). Upon completion, all participants who met the inclusion criteria were randomly assigned to one of three groups (ACT, PP, control group) and received their personal login credentials to the online platform [Synergetic Navigation System, SNS: ccsys.de, Version 3.7.54; 36, 37-39], which was used to administer daily questionnaires and intervention programs. In order to keep the changing societal situation constant for all participants, the study protocol started on April 19th 2020 for all three groups. For a period of 14 days, the two intervention groups received a daily prompt (at 6 AM) via email that their "exercise of the day" was accessible in the SNS. In order to read the exercise instructions, participants had to log into their account via app or web browser. Every day, a new exercise appeared in the system. The intervention period with daily email prompts ended after 14 days.

In the evening (at 5.30 PM), all three groups received an email notification to fill in their daily review questionnaire ("online diary"), every day over the entire study period of 28 days. On day 14, all participants received an email notification to fill in the post measures (t2) available in their SNS account. On day 28, all participants received a notification to fill in the follow-up measures (t3).

Questionnaires and testing material:

At t1 (baseline assessment) participants were asked for information regarding general demographics, their personal living situation, social situation and current status of health. Moreover, participants were asked to indicate the influence of the Corona crisis on their personal lives as well as the adequacy of political measures taken to meet the Corona crisis on visual analogue scales (1 = not at all - 100 = very much).

The following outcome measures were assessed to evaluate the impact of the time spent in relative isolation under conditions of increased stress due to the Corona crisis and potential buffering effects of the interventions: General stress level was assessed using the German version of the stress module of the patient health questionnaire (PHQ-D); as a measure of depression, we used the nine items of the depression module of the patient health questionnaire (PHQ-9); anxiety over the last two weeks was assessed using the 10-item German short version of the State-Trait-Anxiety Inventory (trait version, referenced to the last two weeks); additionally, five items measuring participants' general subjective vitality were included to measure the influence of social distancing on a dynamic feeling of energy and psychosomatic well-being; overall well-being was assessed using five items of the World Health Organization Well-being Index (WHO-5).

"Online diary" and assessment of coping strategies: All participants received a daily review questionnaire which contained two open questions instructing participants to write down 1) relevant events during the day, and 2) things that had helped them in coping positively with the current situation. Participants from the intervention groups were also asked to indicate whether they had carried out the intervention that day (yes/no).

Interventions: see Interventions section

ELIGIBILITY:
Inclusion Criteria:

* knowledge of the German language
* conditions of increased social isolation at the beginning of the study (only individuals were included who were currently staying mostly at home due to the Corona crisis [home office; quarantine measures; stay-at-home orders] with no [or only very few] direct contacts outside of their own household)

Exclusion Criteria:

* acute diagnosis (within the last 3 months) of a mental disorder by a medical professional

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
General stress level (change from baseline/day 1 to post-measurement/day 14) | change from baseline/day 1 to post-measurement/day 14
  General stress level was assessed using the German version of the stress module of the patient health questionnaire (PHQ-). It measures the degree of impairment (not at all, a little, very much; 0-2) in the past four weeks due to nine different sources of stress (assessed by 10 items), such as health worries (item 1), stress due to care issues for family members (item 5), stress at work or in school (item 6), financial concerns (item 7) or having nobody to talk (item 8).
General stress level (change from post-measurement/day 14 to follow-up/day 28) | change from post-measurement/day 14 to follow-up/day 28
  General stress level was assessed using the German version of the stress module of the patient health questionnaire (PHQ-). It measures the degree of impairment (not at all, a little, very much; 0-2) in the past four weeks due to nine different sources of stress (assessed by 10 items), such as health worries (item 1), stress due to care issues for family members (item 5), stress at work or in school (item 6), financial concerns (item 7) or having nobody to talk (item 8).
Symptoms of depression (change from baseline/day 1 to post-measurement/day 14) | change from baseline/day 1 to post-measurement/day 14
  As a measure of depression, we used the nine items of the depression module of the patient health questionnaire (PHQ-9). The instrument assesses impairment (not at all, on some days, more than half of the days, almost every day; 0-3) due to symptoms such as loss of interest and joy in one's activities (item 1) or fatigue and low energy (item 4) over the last two weeks.
Symptoms of depression (change from post-measurement/day 14 to follow-up/day 28) | change from post-measurement/day 14 to follow-up/day 28
  As a measure of depression, we used the nine items of the depression module of the patient health questionnaire (PHQ-9). The instrument assesses impairment (not at all, on some days, more than half of the days, almost every day; 0-3) due to symptoms such as loss of interest and joy in one's activities (item 1) or fatigue and low energy (item 4) over the last two weeks.
Anxiety (change from baseline/day 1 to post-measurement/day 14) | change from baseline/day 1 to post-measurement/day 14
  Anxiety over the last two weeks was assessed using the 10-item German short version of the State-Trait-Anxiety Inventory (trait version, referenced to the last two weeks). The frequency of feelings of calmness (item 3, reversed), lack of self-confidence (item 6), negative thoughts (item 9), feelings of nervousness and unrest (item 10) etc. were rated on an 8-point scale from "almost never" to "almost always" (1-8; due to technical problems, item 7 is missing from this scale).
Anxiety (change from post-measurement/day 14 to follow-up/day 28) | change from post-measurement/day 14 to follow-up/day 28
  Anxiety over the last two weeks was assessed using the 10-item German short version of the State-Trait-Anxiety Inventory (trait version, referenced to the last two weeks). The frequency of feelings of calmness (item 3, reversed), lack of self-confidence (item 6), negative thoughts (item 9), feelings of nervousness and unrest (item 10) etc. were rated on an 8-point scale from "almost never" to "almost always" (1-8; due to technical problems, item 7 is missing from this scale).
Subjective vitality (change from baseline/day 1 to post-measurement/day 14) | change from baseline/day 1 to post-measurement/day 14
  Five items measuring participants' general subjective vitality were included to measure the influence of social distancing on a dynamic feeling of energy and psychosomatic well-being. Participants rated their agreement to statements regarding their general feelings of vitality and aliveness on a 7-point Likert scale from "not at all" to "a lot" (1-7).
Subjective vitality (change from post-measurement/day 14 to follow-up/day 28) | change from post-measurement/day 14 to follow-up/day 28
  Five items measuring participants' general subjective vitality were included to measure the influence of social distancing on a dynamic feeling of energy and psychosomatic well-being. Participants rated their agreement to statements regarding their general feelings of vitality and aliveness on a 7-point Likert scale from "not at all" to "a lot" (1-7).
Overall well-being (change from baseline/day 1 to post-measurement/day 14) | change from baseline/day 1 to post-measurement/day 14
  Overall well-being was assessed using five items of the World Health Organization Well-being Index (WHO-5). Participants needed to determine on a 6-point Likert scale to what extent the items regarding the person's happy mood, calmness, feelings of energy, feelings of recovery in the morning and interest in daily activities had applied during the last two weeks (at no point in time - all the time; 0-5).
Overall well-being (change from post-measurement/day 14 to follow-up/day 28) | change from post-measurement/day 14 to follow-up/day 28
  Overall well-being was assessed using five items of the World Health Organization Well-being Index (WHO-5). Participants needed to determine on a 6-point Likert scale to what extent the items regarding the person's happy mood, calmness, feelings of energy, feelings of recovery in the morning and interest in daily activities had applied during the last two weeks (at no point in time - all the time; 0-5).

SECONDARY OUTCOMES:
Coping strategies | Daily for 14 consecutive days
  All participants received a daily review questionnaire which contained two open questions instructing participants to write down 1) relevant events during the day, and 2) things that had helped them in coping positively with the current situation. From these two questions, we extracted implicit coping strategies.
Daily questionnaire | Daily for 14 consecutive days
  All participants received a daily review questionnaire which contained two open questions (see above) in addition to 20 items assessing: interest and joy during daily activities, nervousness/anxiety, subjective vitality, feelings of optimism, feelings of connectedness, feelings of control (over one's own life), feelings of competency, acceptance of current situation, happiness with the day, physical activity, time spent outside, time spent in the presence of others, time spent virtually with others, structure of the day, influence of the Corona crisis on one's day, stress elicited by the Corona crisis, unhealthy ways of stress regulation, healthy ways of stress regulation, behavior today (adequate - overreacting), feelings of sickness

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Christine Ehlis, PhD, Principal Investigator — University Hospital Tübingen
Locations (1):
- Department of Psychiatry and Psychotherapy, University Hospital Tuebingen, Tübingen, Baden-Wurttemberg, Germany